CLINICAL TRIAL: NCT06303271
Title: Effects of Transcutaneous Auricular Vagus Nerve Stimulation on Dizziness & Balance in Elderly Population With Vestibular Hypofunction
Brief Title: Transcutaneous Auricular Vagus Nerve Stimulation on Dizziness & Balance in Elderly Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MUHAMMAD NISAR
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Vestibular Diseases
Keywords: VNS, Cawthorne exercises
MeSH Terms: conditions — Vestibular Diseases | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vagus Nerve Stimulation (VNS) and Caw Thorne Cooksey (Experimental): Group will receive intervention of 30 minutes daily for 4 weeks (16 sessions).
  Interventions: Other: Vagus Nerve Stimulation (VNS) and Caw Thorne Cooksey
- Caw Thorne Cooksey (Active Comparator): Group will receive intervention of 30 minutes daily for 4 weeks (16 sessions).
  Interventions: Other: Caw Thorne Cooksey

INTERVENTIONS:
Other: Vagus Nerve Stimulation (VNS) and Caw Thorne Cooksey — Study will be conducted after the approval of Ethical review board. After the initial evaluation will be done on participants underlying eligibility criteria. Experimental group will received intervention of 30 minutes daily for 4 weeks (16 sessions). Assessment was done at the baseline, after 2 weeks and after 4 weeks. Intervention Group received non-invasive vagus nerve stimulation at left auricle (because of anatomy of vagus nerve as right VN innervate SA node which is regulating heartbeat and left VN innervates AV node which is responsible for controlling timing of heartbeat) of ear. VNS group received vagus nerve stimulation via Med Fit vagus nerve stimulator at auricle of left ear only as stimulation of right auricular branch of vagus nerve can result in bradycardia. Frequency of stimulation was kept between 15-30Hz. Intensity was gradually increased according to patient's tolerance. The participant was able to withdraw from the trial if he could not tolerate the stimulation
  Arms: Vagus Nerve Stimulation (VNS) and Caw Thorne Cooksey
Other: Caw Thorne Cooksey — Study will be conducted after the approval of Ethical review board. After the initial evaluation will be done on participants underlying eligibility criteria. The control group will intervention of 30 minutes daily for 4 weeks (16 sessions). Caw Thorne Cooksey exercises were carried out during the stimulation of vagus nerve. Although no adverse effects had been reported during the stimulation of left auricular branch of vagus nerve but a pulse oximeter was used during the stimulation to monitor the heart rate.
  Arms: Caw Thorne Cooksey

SUMMARY:
The objective of the study is to determine the effects of transcutaneous auricular vagus nerve stimulation on dizziness and balance on elderly population with unilateral vestibular hypofunction. Patients will be divided into experimental and control group. Randomized participants will be allocated into control and experimental group. Intervention Group A received Vagus Nerve Stimulation (VNS) and Caw Thorne Cooksey exercise while Group group B received Caw Thorne Cooksey exercise only. Both groups received intervention of 30 minutes daily for 4 weeks (16 sessions). Assessment was done at the baseline, after 2 weeks and after 4 weeks

DETAILED DESCRIPTION:
Vestibular hypofunction is also known as vestibulopathy or vestibular dysfunction. It may be unilateral affecting one side or a bilateral vestibulopathy having symptoms on both sides.Typically, vestibular dysfunction results in incapacitating symptoms including imbalance, dizziness, and/or oscillopsia. Symptoms of postural instability and unsteadiness of gait, which aggravate in low light and on uneven terrain, may be given by the patient. The symptoms of the patient may go away while they are sitting or lying still. Without any obvious symptoms, it may be quiet Vestibular hypofunction is a common condition among the elderly population and is associated with a high risk of falls and other balance-related problems. Dizziness and balance problems can significantly impact the quality of life of elderly individuals, leading to a loss of independence and increased risk of injury. Cawthorne Cooksey exercise is a well-established and effective rehabilitation program for individuals with vestibular hypofunction. Transcutaneous auricular vagus nerve stimulation has also been shown to have promising effects on balance and dizziness. However, the combined effect of these two interventions has not been extensively studied.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give consent
2. Age 60 and above
3. Diagnosed patient of unilateral(Left) vestibular hypo function
4. Both Genders
5. BBS with 20-41

Exclusion Criteria:

1. Patient with any neurological impairment (Epilepsy, stroke ALS etc.)
2. Central cause of vestibular hypo function
3. History of vestibular neuritis, concussion, head injury or tumor.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-01-05 (Actual); Study Completion 2025-01-05 (Actual)

PRIMARY OUTCOMES:
The Dix-Hall pike test | 4 weeks
  The Dix-Hall pike test is a test used for diagnosis of BPPV. Therapist must be at side of patient and his/her head is rotated to 45 degree & then therapist suddenly lower the patient in supine lying with 30 degrees below horizontal was the neck's extension. First, the right ear is lowered during the manoeuvre, followed by the left ear. Usually accompanied by vertigo, nystagmus is sought after by the therapist. Nystagmus often lasts 10-20 seconds in BPPV and starts a few seconds later. The patient may experience a brief nystagmus in the opposite direction as they are brought back to an upright posture. When testing is repeated, nystagmus and vertigo usually go down. A test is considered positive by reproduction of vertigo and clinician observation of nystagmus
Berg Balance Scale | 4 weeks
  It consists of 17 items asking patients to rate their responses to statements related to fear of movement and re injury. It has been widely used among patients with various types of pain and has been translated into several languages. The TSK-17 is a useful tool for assessing kinesiophobia and can aid clinicians in developing appropriate treatment plans for patients who may have fear of movement due to pain or injury (20). The TSK exhibit high level of in- ternal consistency across all items and is positively associated with related measures of fear avoidance, pain catastrophizing, pain related disability. In the Finnish version of TSK the test-retest reliability
The Dizziness Handicap Inventory (DHI) | 4 weeks
  The Dizziness Handicap Inventory (DHI) is 25 item self-report questionnaire to asses' vestibular symptom having functional, physical and emotional impact on disability. Patients are asked to answer the questions in Yes, Sometimes and No having 4, 2 and 0 scores. Highest scores are 54+ indicative of severe handicap. Scores b/w 36-52 show moderate and 16-34 means mild handicap.
Dynamic Gait Index (DGI) | 4 weeks
  Dynamic Gait Index (DGI) is another test used for walking balance and is helpful in vestibular problem. DGI is 8 item assessment scale which is scored from 0-3 where 0 is indicative of severe impairment and 3 comes to normal performance. It has total of 24 scores where scores 19 or less indicative of increase risk of falls
Modified Clinical Test of sensory interaction & Balance (MCTSIB) | 4 weeks
  Modified Clinical Test of sensory interaction & Balance (MCTSIB) is used to asses' sensory contribution to postural control and patients attempt to maintain balance. Patients in standing having hand at sides, feet together and perform 4 sensory items like standing on firm surface with eyes open and then close and then on foam surface with eyes open and close and having time of 30 seconds for each activity

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Azhar, MS-NMPT, Principal Investigator — Riphah International University
Locations (1):
- ENT dept. of DHQ Mirpur AJK, Kashmir, Pakistan

IPD SHARING:
Plan to Share IPD: No